CLINICAL TRIAL: NCT00747006
Title: A Phase 2, Single-Center, Open-Label, Pharmacodynamic Clinical Trial to Evaluate the Effect of Technosphere® Insulin Inhalation Powder Safety and Efficacy of Technosphere® Insulin Inhalation Powder (TI Inhalation Powder) Safety and Efficacy of Technosphere® Insulin Inhalation Powder (TI Inhalation Powder) on Postprandial Glucose Levels in Subjects With Type 1 and Type 2 Diabetes Mellitus Ingesting Meals With Varied Carbohydrate Content
Brief Title: Safety and Efficacy of Technosphere® Insulin Inhalation Powder (TI Inhalation Powder)When an Optimal Dose is Taken With Varied Carbohydrate Intake
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-119
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

ARMS (2):
- TI Inhalation Powder (original protocol) (Experimental): Under the original protocol, subjects with Type 1 and Type 2 diabetes will have TI Inhalation Powder administered prandially during dose optimization visits and meal challenge visits (with meals of varying carbohydrate contents). Subjects with Type 2 diabetes will also use TI Inhalation Powder daily at each meal between visits.
  Interventions: Drug: TI Inhalation Powder (original protocol)
- TI Inhalation Powder and Humalog (Amendment 1) (Other): Under Amendment 1, TI Inhalation Powder will be administered prandially to a new subset of subjects with Type 2 diabetes during TI dose optimization visits and TI meal challenge visits (with meals of varying carbohydrate contents). Subjects will be crossed over to administration of Humalog 15 minutes before meals during Humalog dose optimization visits and Humalog meal challenge visits (with meals of varying carbohydrate contents). Subjects will also use TI Inhalation Powder daily at each meal between visits.
  Interventions: Drug: TI Inhalation Powder and Humalog (Amendment 1)

INTERVENTIONS:
Drug: TI Inhalation Powder and Humalog (Amendment 1) — Subcutaneous (sc) rapid acting analog to be administered at one half of the meal challenge visits 15 minutes before a meal. Only the last 5 - 10 patients (Type 2) will be undergoing this amendment to the protocol.
  Arms: TI Inhalation Powder and Humalog (Amendment 1)
Drug: TI Inhalation Powder (original protocol) — Inhaled insulin technology to be administered immediately before a meal (prandially) for glucose control in Type 1 or Type 2 diabetics
  Arms: TI Inhalation Powder (original protocol)

SUMMARY:
The purpose of this study is to determine if, once a favorable dose of TI Inhalation Powder is established for either a type 1 or 2 patient, based on a average diabetic meal, the patient's favorable dose can be used safely, regardless of change in meal carbohydrate content. Patients were randomly assigned to various carbohydrate loads (0%, 50%, 100%, 150% or 200%). The 100% carbohydrate load was determined based upon their standard insulin dose for their normal meal.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses of type 1 or type 2 diabetes mellitus
* Fasting Plasma Glucose (FPG) 80, 140 mg/dL and glycated hemoglobin (A1C) > 6.5% and < or = 10.0%.
* Body mass index (BMI) of < or = 40 kg/m2
* Non-smokers (never smoked or former smokers [= 6 months since cessation]) and a urine cotinine level < or = 100 ng/dL
* Forced expiratory volume in 1 second (FEV1) = 70% Third National Health and Nutrition Examination Survey (NHANES III) Predicted; pre-bronchodilator FEV1 as a percentage of forced vital capacity (FEV1/Forced vital capacity(FVC)) = 70%
* For subjects with type 2 diabetes mellitus: Currently receiving oral diabetic treatment or basal insulin +/- oral diabetic treatment

Exclusion Criteria:

* History of chronic obstructive pulmonary disease (COPD), clinically proven asthma, and/or any other clinically important pulmonary disease confirmed by pulmonary function test (PFT) and/or radiologic findings
* Elevated liver function test (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3 times the normal reference range or bilirubin > 1.5 times the reference range)
* Previous use of Exubera; use of Symlin (pramlintide acetate) and/or Byetta (exenatide) within the past 12 weeks
* Unstable diabetes control and evidence of severe complications of diabetes mellitus (ie, autonomic neuropathy)
* Exposure to any investigational product(s) in the past 12 weeks
* For subjects with type 2 diabetes mellitus: In subjects taking metformin, serum creatinine > 1.4 mg/dL in female subjects and > 1.5 mg/dL in male subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sansum Medical Research Institute, Santa Barbara, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Original Protocol Type 1 Diabetes: Original protocol participants with Type 1 diabetes given Technosphere Insulin (TI - doses individualized for each patient) at various carbohydrate loads [0%, 50%, 100% (reference), 200%, and if necessary, 150%)
- Original Protocol Type 2 Diabetes: Original protocol participants with Type 2 diabetes given Technosphere Insulin (TI - doses individualized for each patient) at various carbohydrate loads [0%, 50%, 100% (reference), 200%, and if necessary, 150%)
- Amendment 1 Type 2 Diabetes: Protocol amendment 1 participants with Type 2 diabetes given humalog (doses individualized for each patient) or Technosphere Insulin (doses individualized for each patient) at various carbohydrate loads [0%, 50%, 100% (reference), 200%, and if necessary, 150%)
Period: Overall Study
Arm/Group | Original Protocol Type 1 Diabetes | Original Protocol Type 2 Diabetes | Amendment 1 Type 2 Diabetes
Started | 7 | 8 | 3
Completed | 4 | 7 | 2
Not Completed | 3 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Subjects. Patients were randomly assigned to various carbohydrate loads (0%, 50%, 100%, 150% or 200%). The 100% carbohydrate load was determined based upon their standard insulin dose for their normal meal.
Groups:
- Total: Total of all reporting groups
Arm/Group | Original Protocol Type 1 Diabetes | Original Protocol Type 2 Diabetes | Amendment 1 Type 2 Diabetes | Total
Number analyzed (Participants) | 7 | 8 | 3 | 18
Age, Continuous [Mean (Full Range); unit: years] | 40.7 [18 to 54] | 59.4 [50 to 70] | 50.7 [48 to 52] | 50.7 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 5 | 7 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Lunch Plasma Glucose Time 0 Corrected AUC (0-240) - Original Protocol (TI Treated Type 1 Subjects)
Description: AUC (area under the plasma glucose - time curve) from time 0 (immediately before starting meal) to 240 minutes after the start of the meal when the curve is above time 0 value.
  AOC (area over the plasma glucose - time curve) from time 0 (immediately before starting meal) to 240 minutes after the start of the meal when the curve is below time 0 value.
  TIme 0 corrected AUC (0-240) = AUC - AOC
Time Frame: 0 to 240 minutes
Population: Original Protocol Type 1 Diabetes Mellitus Technosphere Insulin Treated; 50% carbohydrate load was administered but not completed due to all subjects having hypoglycemia, 0% carbohydrate load was deemed unsafe by PI
Measure: Mean (Full Range); unit: min*mg/dL
Groups:
- 100% Carbohydrate Load: Standard meal to which subjects titrated their insulin dose.
- 0% Carbohydrate Load: Fasting state
- 50% Carbohydrate Load: Meal consisting of half of the carbohydrates from the standard meal
- 150% Carbohydrate Load: Meal consisting of 1.5 times the carbohydrate load of the standard meal.
- 200% Carbohydrate Load: Meal consisting of 2 times the carbohydrate load of the standard meal.
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
min*mg/dL | -41.44 [-43.44 to -39.43] |  |  | 251.65 [24.08 to 490.63] | 454.07 [329.64 to 636.50]

2. Primary Outcome: Breakfast Plasma Glucose Time 0 Corrected AUC(0-240) - Original Protocol (TI Treated Type 1 Subjects)
Description: as for outcome 1
Time Frame: 0 to 240 minutes
Population: Original Protocol Type 1 Diabetes Mellitus Technosphere Insulin Treated; 0% carbohydrate load was deemed unsafe by PI
Measure: Mean (Full Range); unit: min*mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 0 | 3 | 2 | 3
min*mg/dL | 104.32 [14.50 to 194.13] |  | 10.80 [-44.86 to 98.50] | 199.35 [116.70 to 282.00] | 440.90 [269.18 to 583.13]

3. Primary Outcome: Lunch Plasma Glucose Time 0 Corrected AUC(0-240) - Amendment 1 (TI Treated Type 2 Subjects)
Description: as for outcome 1
Time Frame: 0 to 240 minutes
Population: Protocol Amendment 1 Type 2 Diabetes Mellitus Technosphere Insulin Treated Subjects; 150% carbohydrate load was not done per protocol since the 200% carbohydrate load was administered
Measure: Mean (Full Range); unit: min*mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 2
min*mg/dL | -6.11 [-22.63 to 10.41] | -74.26 [-99.88 to -48.63] | -22.80 [-22.80 to -22.80] |  | 11.56 [-2.36 to 25.47]

4. Primary Outcome: Lunch Plasma Glucose Time 0 Corrected AUC(0-240) - Amendment 1 (Humalog Treated Type 2 Subjects)
Description: as for outcome 1
Time Frame: 0 to 240 minutes
Population: Protocol Amendment 1 Type 2 Diabetes Mellitus Humalog Treated Subjects; 150% carbohydrate load was not done per protocol since the 200% carbohydrate load was administered
Measure: Mean (Full Range); unit: min*mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 2 | 2 | 0 | 2
min*mg/dL | 15.77 [9.48 to 22.06] | -51.26 [-89.13 to -13.38] | 4.18 [-15.39 to 23.75] |  | -8.15 [-68.76 to 52.47]

5. Primary Outcome: Lunch Plasma Glucose Excursion - Original Protocol (TI Treated Type 1 Subjects)
Description: Excursion is the difference between plasma glucose Cmax and Cmin (Cmax - Cmin) at lunch
Time Frame: 0 to 240 minutes
Population: as for outcome 1
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
mg/dL | 54.00 [42.00 to 66.00] |  |  | 129.67 [75.00 to 210.00] | 201.00 [163.00 to 231.00]

6. Primary Outcome: Breakfast Plasma Glucose Excursion - Original Protocol (TI Treated - Type 1 Subjects)
Description: Excursion is the difference between plasma glucose Cmax and Cmin (Cmax - Cmin) at breakfast
Time Frame: 0 to 240 minutes
Population: Original Protocol Type 1 Diabetes Mellitus Technosphere Insulin Treated; 0% carbohydrate load was deemed unsafe by PI
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 0 | 3 | 2 | 3
mg/dL | 53.50 [43.00 to 64.00] |  | 44.33 [42.00 to 48.00] | 89.50 [78.00 to 101.00] | 186.33 [134.00 to 234.00]

7. Primary Outcome: Lunch Plasma Glucose Excursion - Amendment 1 ( TI Treated Type 2 Subjects)
Description: Excursion is the difference between plasma glucose Cmax and Cmin (Cmax-Cmin) at lunch
Time Frame: 0 to 240 minutes
Population: Protocol Amendment 1 Type 2 Diabetes Mellitus TI Treated Subjects; 150% carbohydrate load was not done per protocol since the 200% carbohydrate load was administered
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 2
mg/dL | 29.50 [26.00 to 33.00] | 14.50 [13.00 to 16.00] | 16.00 [16.00 to 16.00] |  | 18.50 [17.00 to 20.00]

8. Primary Outcome: Lunch Plasma Glucose Excursion - Amendment 1 (Humalog Treated Type 2 Subjects)
Description: Excursion is the difference between plasma glucose Cmax and Cmin (Cmax-Cmin) at lunch
Time Frame: 0 to 240 minutes
Population: as for outcome 4
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 2 | 2 | 0 | 2
mg/dL | 44.50 [44.00 to 45.00] | 20.00 [9.00 to 31.00] | 23.50 [11.00 to 36.00] |  | 45.50 [35.00 to 56.00]

9. Secondary Outcome: Lunch Plasma Glucose AOC (0-240) - Original Protocol (TI Treated Type 1 Subjects)
Description: Area over the plasma glucose - time curve from time 0 (immediately before starting lunch) to 240 minutes after the start of the lunch
Time Frame: 0 to 240 minutes
Population: as for outcome 1
Measure: Mean (Full Range); unit: min*mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 0 | 0 | 3 | 3
min*mg/dL | 53.89 [47.61 to 60.16] |  |  | 19.16 [0.00 to 57.49] | 8.77 [0.00 to 26.05]

10. Secondary Outcome: Breakfast Plasma Glucose AOC(0-240) - Original Protocol (TI Treated Type 1 Subjects)
Description: Breakfast area over the plasma glucose - time curve from time 0 (immediately before breakfast) to 240 minutes after start of breakfast
Time Frame: 0 to 240 minutes
Population: Original Protocol Type 1 Diabetes Mellitus Technosphere Insulin Treated; 0% carbohydrate load was deemed unsafe by PI
Measure: Mean (Full Range); unit: min*mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 0 | 3 | 2 | 3
min*mg/dL | 10.25 [0.00 to 20.50] |  | 30.45 [0.00 to 59.00] | 6.30 [0.00 to 12.60] | 3.18 [0.00 to 9.55]

11. Secondary Outcome: Lunch Plasma Glucose AOC(0-240) - Amendment 1 (TI Treated Type 2 Subjects)
Description: Lunch area over the plasma glucose - time curve from time 0 (immediately before breakfast) to 240 minutes after start of lunch
Time Frame: 0 to 240 minutes
Population: as for outcome 3
Measure: Mean (Full Range); unit: min*mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 2 | 1 | 0 | 2
min*mg/dL | 18.00 [5.36 to 30.63] | 74.26 [48.63 to 99.88] | 24.04 [24.04 to 24.04] |  | 5.65 [1.53 to 9.77]

12. Secondary Outcome: Lunch Plasma Glucose AOC(0-240) - Amendment 1 (Humalog Treated Type 2 Subjects)
Description: as for outcome 11
Time Frame: 0 to 240 minutes
Population: as for outcome 4
Measure: Mean (Full Range); unit: min*mg/dL
Arm/Group | 100% Carbohydrate Load | 0% Carbohydrate Load | 50% Carbohydrate Load | 150% Carbohydrate Load | 200% Carbohydrate Load
Number analyzed (Participants) | 2 | 2 | 2 | 0 | 2
min*mg/dL | 14.60 [11.34 to 17.86] | 51.63 [14.13 to 89.13] | 12.52 [7.50 to 17.53] |  | 40.84 [10.89 to 70.79]

ADVERSE EVENTS:
Groups:
- TI Original Protocol Type 1 DM: Original protocol type 1 diabetes mellitus subjects
- TI Original Protocol Type 2 DM: Original protocol type 2 diabetes mellitus subjects
- TI Amendment 1 Type 2 DM: Technosphere Insulin treated subjects in protocol amendment 1
- Humalog Amendment 1 Type 2 DM: Humalog treated subjects in protocol amendment 1
Arm/Group | TI Original Protocol Type 1 DM | TI Original Protocol Type 2 DM | TI Amendment 1 Type 2 DM | Humalog Amendment 1 Type 2 DM
Serious Adverse Events (participants affected / at risk) | 0/7 | 3/8 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 7/7 | 7/8 | 3/3 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TI Original Protocol Type 1 DM (N=7) | TI Original Protocol Type 2 DM (N=8) | TI Amendment 1 Type 2 DM (N=3) | Humalog Amendment 1 Type 2 DM (N=2)
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Renal papillary necrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TI Original Protocol Type 1 DM (N=7) | TI Original Protocol Type 2 DM (N=8) | TI Amendment 1 Type 2 DM (N=3) | Humalog Amendment 1 Type 2 DM (N=2)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 6 | 2 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Venipuncture site thrombosis (General disorders) | 1 | 0 | 0 | 0
Allergy to plants (Immune system disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
- Early termination of trial leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.